CLINICAL TRIAL: NCT04867720
Title: Multi-center, Single Arm, Open-label, Phase 4 STudy to Evaluate the Efficacy and Safety of CertiroBELL® Tablet Plus TAcrolimus in Primary Living Donor Liver Transplant Recipients
Brief Title: Efficacy and Safety of CertiroBell® Tablet Plus Tacrolimus in Primary Living Donor Liver Transplant Recipients
Acronym: STELLA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B95_03LT2001
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Liver Transplant
Keywords: Everolimus; CertiroBell; Tacrolimus
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CertiroBell Tablet (Experimental): Use in combination with Tacrolimus at least 6 months after liver transplantation.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — - Oral intake, BID - After first dose 1mg(total 2mg daily), check the blood concentration of everolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 3~8mg/mL.
  Other Names: CertiroBell Tab.

SUMMARY:
To evaluate the efficacy and safety of CertiroBell® tablet plus tacrolimus

DETAILED DESCRIPTION:
This study is multi-center, single arm, open-label, phase 4 study to evaluate the efficacy and safety of CertiroBell® tablet plus tacrolimus in primary living donor liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had liver transplantation from living donor and had passed over 3 months since operation.
2. Over 20 years old
3. Patients who are being treated with Tacrolimus at screening visit
4. Patients who agreed to written informed consent

Exclusion Criteria:

1. Patients who had received non-liver organs before liver transplantation or had received other organs while receiving liver.
2. Patients who had auxiliary partial orthotopic liver transplantation or had bioartifical liver
3. Patients who have been diagnosed with acute rejection within 6 months and have been treated
4. Patients who had hepatic artery complication such as hepatic artery thrombosis within recent 6 months
5. Patients who have been diagnosed with malignant tumor within 5 years(however, the following will be excepted)

   * fully recovered from skin cancer(squamous cell/basal cell carcinoma or thyroid cancer)
   * haptocellular carcinoma without main vessel invasion
6. Patients with severe systemic infection
7. Patients who are difficult to communicate due to mental disorder
8. Patients who are in treatment for hapatitis, or are over 3 times higher than upper normal limit in liver function test(T-bilirubin, AST, ALT) or over 5 times higher than normal limit of ALP
9. Patients who are(at screening visit)

   * WBC<1,500/mm^3
   * PLT<30,000/mm^3
   * over 1.0 in Protein/creatinine ratio(UA test)
   * eGFR<30mL/min/1.73m^2(MDRD)
   * Total Cholesterol>350mg/dL or Triglycerides>500mg/dL
10. Patients taking HCV(hapatitis C virus) therapeutic drug or anti-HCV positive patients who have positive result in HCV RNA test at screening visit
11. Patients who had plasmapheresis within 1 week
12. Those who are pregnant, nursing, or are not practicing contraception with appropriate method
13. Patients who had plasmapheresis within 3 months
14. if participated in other trail within 4 weeks(28 days)
15. In investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-10-10 (Estimated); Study Completion 2023-02-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure | until 24 weeks after taking medicine
  composite efficacy failure include biopsy-confirmed acute rejection, graft loss, death, or follow-up failure

SECONDARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection | until 24 weeks after taking medicine
  acute rejection confirmed by result of biopsy(over 4 points of RAI score)
Pathological result, time of occurrence, treatment method and treatment result of acute rejection confirmed by biopsy(over 4 points of RAI score) | until 24 weeks after taking medicine
  details of acute rejection confiremd by result of biopsy(over 4 points of RAI score)
Survival rate of patients | until 24 weeks after taking medicine
  Survival rate of patients
Survival rate of transplanted organ | until 24 weeks after taking medicine
  Survival rate of transplanted organ
Incidence rate of liver cancer | until 24 weeks after taking medicine
  Incidence rate of liver cancer
Recurrence rate of liver cancer | until 24 weeks after taking medicine
  Recurrence rate of liver cancer
Incidence rate of CMV infection | until 24 weeks after taking medicine
  Incidence rate of CMV infection
Variation of serum creatinine, eGFR(estimated glomerular filtration rate) compared to baseline using MDRD(Modification of Diet in Renal Disease) | until 24 weeks after taking medicine
  eGRF using MDRD(Modification of Diet in Renal Disease) method

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Suk Suh, M.D., Ph.D., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hosipital, Seoul, South Korea